CLINICAL TRIAL: NCT03289507
Title: Longvida Curcumin Human Pharmacokinetics (PK) Study
Brief Title: Longvida Curcumin Human Pharmacokinetics Study
Acronym: CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Verdure Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB2017-086
Record Dates: First submitted 2017-09-14; First posted 2017-09-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Longvida Curcumin; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment1 (Active Comparator): Longvida Capsule formulation A
  Interventions: Dietary Supplement: Treatment1
- Treatment 2 (Active Comparator): Longvida Capsule formulation B
  Interventions: Dietary Supplement: Treatment2
- Treatment3 (Experimental): Curcuma longa extract of Rhizomes
  Interventions: Dietary Supplement: Treatment3

INTERVENTIONS:
Dietary Supplement: Treatment1 — Longvida Capsule formulation A
  Arms: Treatment1
Dietary Supplement: Treatment2 — Longvida Capsule formulation B
  Arms: Treatment 2
Dietary Supplement: Treatment3 — Curcuma longa extract of Rhizomes
  Arms: Treatment3

SUMMARY:
The primary objective of the study is to characterize the curcumin metabolites of 2 different capsule formulations of curcumin relative to unformulated Curcuma longa extract of Rhizomes including assessing relative bioavailability and absorption/kinetic profile of curcumonoids and their metabolites in human plasma and urine after acute consumption.

DETAILED DESCRIPTION:
This study is a randomized, 3-arm, double-blinded, within subject cross-over trial focused on understanding pharmacokinetic profile of curcuminoids and their metabolites after intake of curcumin supplement with different capsule formulations.

A planned sample size of 6 will be enrolled into the study. This study will require one initial screening visit and 3 weekly visits. This study will take approximately 4 weeks per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, subjects will be invited to participate in the study for 3 study days. Subjects will be instructed to maintain their usual diet pattern and physical activity throughout study duration.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed health Care Professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Subjects will be randomized to receive a curcumin supplement based on randomized treatment sequences for 3 study visits immediately after fasting blood draw. The sequences of receiving the supplement at each visit will be randomly assigned based on treatment sequences.

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.5, 1, 2, 4, 6, and 8 hour (h) for assessment of change in plasma curcuminoids and metabolites. A standard breakfast will be provided immediately after the 0.5 h blood collection and standard lunch after 6 h blood collection. Urine samples will be collected at 0 (fasting), 4 and 8 h.

ELIGIBILITY:
Inclusion Criteria:

* • Men or women, 20-45 years of age with body mass index (BMI) in range from 18.5 to 24.9 kg/m2

  * Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 2 years)
  * No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease that may interfere with study outcomes
  * Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, gastrointestinal medications, antibiotics, anti-inflammatory drugs, dietary supplements including fiber supplements, prebiotics and probiotics, etc.
  * Able to provide informed consent
  * Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, blood and urine sample collection procedures and study visit schedule)
  * Minimum weight of 45 kg

Exclusion Criteria:

* Men and women who smoke

  * Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
  * Men and women known to have/diagnosed with diabetes mellitus
  * Men and women who have fasting blood glucose concentrations > 125 mg/dL
  * Men and women who have uncontrolled blood pressure >160 mmHg (systolic) or 100 mmHg (diastolic)
  * Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
  * Men and women with cancer other than non-melanoma skin cancer in previous 5 years
  * Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
  * Women who are known to be pregnant (pregnancy test will be completed for female subjects) or who are intending to become pregnant over the course of the study
  * Women who are lactating
  * Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
  * Men and women who has participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
  * Men and women who have donated blood within 3 months of the Screening Visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
  * Men and women who are vegans
  * History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
  * Substance (alcohol or drug) abuse within the last 2 years
  * Excessive coffee and tea consumers (> 5 cups/day)
  * Men and women who do excessive exercise regularly or athlete
  * Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
  * Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
  * Unusual working hours i.e., working overnight (e.g. 3rd shift)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in plasma curcumin metabolites among 3 different treatments | 8 hours Postprandial Study
  Differences in plasma metabolites among 3 treatments

SECONDARY OUTCOMES:
Changes in urine metabolites among 3 different treatments | 8 hours Postprandial Study
  Differences in urine metabolites among 3 treatments

CONTACTS AND LOCATIONS:
Overall Officials: Britt M Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States